CLINICAL TRIAL: NCT01578460
Title: Healthy Moms, Healthy Babies: A Strategy to Improve the Care and OUtcome of Diabetes in Pregnancy in On-Reserve First Nations Women
Brief Title: Healthy Moms, Healthy Babies
Acronym: HMHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stewart Harris (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Stewart Harris, Professor, CDA Chair in Diabetes Management, Ian McWhinney Chair of Family Medicine Studies, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R-11-223; 17686 (Other: Research Ethics Board)
Record Dates: First submitted 2012-04-05; First posted 2012-04-17 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus; Gestational Diabetes
Keywords: Pregnancy; Gestational Diabetes; Type 2 Diabetes Mellitus; Continuous Glucose Monitor; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Participants will self-select which group they wish to participate in at time of consent. The control group will use standard glucose meter testing to monitor their glucose levels.
  Interventions: Device: Glucose Meter
- Continuous Glucose Monitor (CGM) Group (Experimental): Participants will self-select which group they wish to participate in at time of consent. The CGM group will utilize the iPro2 CGM to monitor their glucose levels during their 28, 32, and 36 week of gestation.
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Participants in the CGM group will be asked to monitor their blood glucose for 5 days for the 28th, 32nd and 36th week of gestation using the iPro2 CGM.
  Other Names: iPro2 by Medtronic
  Arms: Continuous Glucose Monitor (CGM) Group
Device: Glucose Meter — Participants in the control group will be asked to monitor their blood glucose for 5 days for the 28th, 32nd and 36th week of gestation using a glucose meter.
  Other Names: Lifescan One Touch Ultra Mini
  Arms: Control Group

SUMMARY:
Poor glucose control during pregnancy is a significant concern for Canadian women with diabetes. This problem is magnified in First Nations women, who have among the highest rates of gestational diabetes (GDM) in the world (up to 18% of First Nations women will develop GDM during pregnancy and 70% of these will go on to develop type 2 diabetes later). Continuous glucose monitoring (CGM) technology has the potential to help women maintain tighter control during pregnancy, however, in the First Nations population, there are many unique barriers that may affect use of this technology. Such barriers include remoteness of the community, cultural apprehension, lack or difficulty of access to care, and language differences.

A total of 60 participants from three participating First Nations communities in Southern Ontario will participate in the study. Participants will self-select to either the CGM group (n=30) or the control group (n=30) after consenting to participate in the study. Participants in both groups will be asked to monitor their blood glucose for 5 days for the 28th, 32nd and 36th week of gestation. Primary outcomes to be evaluated include maternal A1c and offspring birth weight. To assess the feasibility and acceptability of CGMs among First Nations women, a questionnaire will be distributed to participants to gather insight into their rationale for enrolling into either group. Recruitment rates for both groups will also be used to assess feasibility and acceptability of CGMs. Additionally, all participants will be encouraged to participate in a community lifestyle program consisting of 30-min exercise sessions offered five days a week. The community lifestyle program will be adapted to the community, linked to existing programs with support from program personnel and will include educational sessions related to diabetes and healthy lifestyles. It is hypothesized that through participation in the community lifestyle program, pregnant First Nations women with diabetes will experience a decrease in their blood glucose values post-exercise, mitigate excessive weight gain and normalize their A1c's. It is further hypothesized that an increase in women's regular physical activity levels, the number of steps taken and knowledge of diabetes will be observed.

ELIGIBILITY:
Inclusion Criteria:

* First Nations (self-identified)
* On-reserve (living or receiving care)
* Informed consent to participate
* Adults aged 18 years or older
* Diagnosed with gestational diabetes (GDM) or type 2 diabetes (T2DM)
* Pregnant (less than or equal to 36 weeks o gestation)
* Consent to have primary care giver informed of participation in teh project
* Willingness to perform required study and data collectin procedures and adhere to the operating requirements of the iPro2 and/or the glucose meter
* Willingness to wear the iPro 2 continuous glucose monitor (CGM) for 5 days for the 28th, 32nd, 36th week of pregnancy (for participants in the CGM group)
* Willingness to perform at least 4 finger prick testing per day during the Monitoring Week of the 28th, 32nd, 36th week of pregnancy (for CGM and control group)

Exclusion Criteria:

* Lack of decision making capacity to provide consent
* Participating in another diabetes and/or lifestyle improvement research project
* Non-First Nations descent
* Pregnant diagnosed with type 1 diabetes
* Pregnant not diagnosed with GDM or T2DM
* Pregnant women past 36th week of gestation
* Participants who do not consent to have their primary care giver informed of project participation
* The participant has a history of tape allergies that have not been resolved
* The participant has any skin abnormality (e.g. Psoriasis, rash, staphylococcus infection) that has not been resolved and would inhibit her from wearing the sensor
* Any other condition (s) that in the Investigator's opinion would warrant exclusion from the study or prevent the participant from completing the project

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-08-29 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
Maternal HbA1c | 24, 28, 32 and 36th week of gestation. This will occur between May 2012 to September 2014
  Lab collected at the specific time periods listed above.
Offspring Birth Weight | At Delivery. This will occur between May 2012 to September 2014.
  Offspring birth weight will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.

SECONDARY OUTCOMES:
1 hour post-prandial glucose measurements (maternal) | 28, 32 and 36th week of gestation. This will occur between May 2012 to September 2014.
  This will be collected from the CGM or glucose meter, depending on the group the participant consents to take part in.
Weight gain (maternal) | Weight is recorded at each visit from May 2012 to September 2014.
  Baseline weight is collected from Antenatal Record 1 and 2 (Ontario Ministry of Health and Long-Term Care forms). Follow-up weight measurements are done at each visit until delivery. Weight gain is calculated from the baseline and follow-up measurements.
Maternal diabetes treatment | 28, 32, and 36 weeks of gestation. This will occur between May 2012 to September 2014.
  Baseline treatment will be collected from Antenatal Record 1 and 2 (Ontario Ministry of Health and Long-Term Care forms) if available.
Daily mean glucose values (maternal) | 28, 32 and 36th week of gestation. This will occur between May 2012 to September 2014.
  This will be calculated from the glucose measurements taken using either the CGM or the glucose meter.
Insulin Use (maternal) | 24, 28, 32, and 36 weeks of gestation. This will occur between May 2012 to September 2014.
  Baseline insulin use will be collected from Antenatal Record 1 and 2 (Ontario Ministry of Health and Long-Term Care forms) if available.
Neonatal gestational age | At Delivery. This will occur between May 2012 to September 2014.
  Neonatal gestational age will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Neonatal hypoglycemia | At Delivery. This will occur between May 2012 to September 2013.
  Neonatal hypoglycemia will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Neonatal Intensive Care Unit (NICU) Admission | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Number of days in the hospital (neonatal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Birth injuries (neonatal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Jaundice (neonatal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Delivery in a community or teaching hospital | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Caesarean section rate (maternal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal Discharge Summary.
Delivery Methods | At Delivery. This will occur between May 2012 to September 2014.
  Forceps, vacuum-assisted. This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Cephalopelvic disproportion | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.
Number of days in hospital post delivery (maternal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Maternal Discharge Summary.
Shoulder Dystocia (neonatal) | At Delivery. This will occur between May 2012 to September 2014.
  This will be collected from the Neonatal Examination Form/Birth Record and Maternal and Offspring Discharge Summaries.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Harris, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Western University, London, Ontario, Canada